CLINICAL TRIAL: NCT06611293
Title: HOspital Versus Primary Care Breath Test Environment (HOPE) Study
Acronym: HOPE
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 24HH8812
Record Dates: First submitted 2024-09-16; First posted 2024-09-24 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Breath Test
MeSH Terms: interventions — Breath Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Volunteers taking part in study
  Interventions: Diagnostic Test: Breath test

INTERVENTIONS:
Diagnostic Test: Breath test — Participants will perform breath testing in Primary care followed by Secondary care on Day 1. At each location, participants will be asked to perform three breath tests (15 minutes apart). The environmental air will also be sampled.
  This entire process will be repeated in the reverse order (i.e. breath testing in Secondary care followed by Primary care on Day 2).
  Participants will be asked to maintain a clear fluid diet for a minimum of six hours prior to breath collection on both Day 1 and Day 2 of sampling.

SUMMARY:
Through the HOPE study, the intention would be to determine whether exhaled breath volatile organic compound (VOC) profiles in Primary care differ from Secondary care. The intention would also be to assess intra-subject variability of participants. This would allow us to determine if the results of breath samples are reproducible regardless of whether they are performed in a Primary or Secondary care environment. This would support the clinical translation of breath research outcomes from studies performed in Secondary care, despite the breath test being intended for use in Primary care.

The chief investigator of the HOPE study is Professor George Hanna (Head of Department of Surgery and Cancer, and Professor of Surgical Sciences at Imperial College London).

DETAILED DESCRIPTION:
A breath test is a non-invasive investigation. The use of a breath test as a triage tool - for cancer or other diseases - in symptomatic patients could identify high-risk patients who should be referred for investigations at an earlier stage. This would increase the proportion of appropriate referrals from Primary care and improve adherence to National Institute for Clinical Health and Excellence (NICE) guidance. If a General Practitioner (GP) is presented with a patient with symptoms that do not prompt referral under NICE guidelines, he/she would no longer need to watch-and-wait to see if their symptoms worsen, but could instead offer a breath test immediately. Breath samples would be collected and sent to a regional laboratory for analysis. A positive result would warrant immediate referral for further specialised investigations, whilst a negative test would permit the GP to reassure the patient and offer re-testing if symptoms persist.

The MAGIC (Methodological Approaches towards a GastroIntestinal Cancer test) study was performed to assess whether breath testing is feasible in Primary care. In this study, 1002 patients took part in the breath test in Primary care. Ninety-nine percent of patients found the breath test very easy or easy to perform, and it was demonstrated that breath testing is feasible in Primary care.

However, the potential for an individual's exhaled breath VOC profile to change when measured across Primary and Secondary care sites has not yet been investigated.

ELIGIBILITY:
Inclusion Criteria:

Participants will be:

* Aged ≥ 18 years old
* Willing and able to provide informed consent to take part in study.

Exclusion Criteria:

* Pregnant women will be excluded from this study. With the exception of pregnant women, there are no additional strict exclusion criteria as individuals will act as their own control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Volunteers will be recruited to provide breath samples in both Primary and Secondary Care environments.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
The variation in exhaled breath VOC profile in the participants in Primary versus Secondary Care setting. | 2 years
  An exploratory analysis will be performed to identify and exclude contaminated samples. Linear mixed models will be fitted for each compound's measurements to estimate components of variation (between individuals, occasions and repeat samples), and confirm that there is no effect of ordering (hospital-GP vs GP-hospital). Repeatability of each day-location combination will be summarised as the intra-class correlation coefficient (ICC) and the coefficient of variation (CV).
  The observed differences will be compared with the clinically acceptable limits for each VOC to identify the proportion of GP-hospital differences that fall within these limits. For each VOC, the ICC, CV and the limits of agreement with 95% confidence interval will be reported, along with how they compare with the clinically acceptable differences.

SECONDARY OUTCOMES:
The intra-subject variability in exhaled breath VOCs when breath is sampled 15 minutes apart on different days. | 2 years
  Please see "Description" for "Primary Outcome Measure".

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London, London, United Kingdom